CLINICAL TRIAL: NCT01908972
Title: The Safety and Efficiency of Propranolol as an Initial Treatment for Pediatric Hemangioma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12172-MM-231
Record Dates: First submitted 2013-07-09; First posted 2013-07-26 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2016-02

CONDITIONS: Hemangioma
Keywords: Hemangioma; Propranolol; prednisolone; steroid
MeSH Terms: conditions — Hemangioma | interventions — Prednisolone; Steroids; Propranolol; Adrenergic beta-Antagonists

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisolone (Active Comparator): Patients who will receive prednisolone medication (2 mg/kg/day ) for 16 weeks
  Interventions: Drug: Prednisolone
- Propranolol (Experimental): Patients who will receive propranolol medication 2 mg/kg/day for 16 weeks
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Prednisolone — 2mg/kg/day for 16weeks
  Other Names: steroid
  Arms: Prednisolone
Drug: Propranolol — 2mg/kg/day for 16weeks
  Other Names: beta-blocker
  Arms: Propranolol

SUMMARY:
The purpose of this study is to determine the safety and efficiency of Propranolol as an initial treatment for pediatric hemangioma.

DETAILED DESCRIPTION:
* Randomized (A group : propranolol, B group : prednisolone)
* A group : 3 days admission and medication for 16 weeks
* B group : medication for 16 weeks without admission
* Hemangioma volume comparison by using MRI
* other measurement and drug adverse reaction monitoring

ELIGIBILITY:
Inclusion Criteria:

* Hemangioma patient ( 0 ~ 9 months old)
* No treatment before
* 10 ~ 20 % volume increase in 2 ~ 4 weeks
* Hemangioma that caused organ function
* Hemangioma that will cause aesthetic problem

Exclusion Criteria:

* Cardiovascular disease (impossible to use propranolol)
* Drug adverse reaction or allergy history (propranolol, steroid)
* Bradycardia, Atrioventricular block, atrial block
* Cardiogenic Shock
* Right heart failure (pulmonary hypertension)
* Congestive heart failure
* Hypotension
* Peripheral nerve disease (moderate)
* Angina
* Hormone deficiency patient
* Pulmonary disease (asthma)
* diabetic ketoacidosis
* laser treatment history

Max Age: 9 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2013-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-Duk Park, MD, Ph D, Study Director — Seoul National University Hospital; Tae Hyun Choi, MD, Ph D, Study Director — Seoul National University Hospital
Locations (1):
- Seould National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kim KH, Choi TH, Choi Y, Park YW, Hong KY, Kim DY, Choe YS, Lee H, Cheon JE, Park JB, Park KD, Kang HJ, Shin HY, Jeong JH. Comparison of Efficacy and Safety Between Propranolol and Steroid for Infantile Hemangioma: A Randomized Clinical Trial. JAMA Dermatol. 2017 Jun 1;153(6):529-536. doi: 10.1001/jamadermatol.2017.0250. PMID 28423174

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prednisolone | Propranolol
Started | 17 | 17
Completed | 15 | 17
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prednisolone | Propranolol | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 17 | 34
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: months] | 3.0 [0.8 to 8.0] | 3.6 [0.3 to 8.2] | 3.3 [0.3 to 8.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 17 | 17 | 34
Hemangioma volume by MRI [Mean (Standard Deviation); unit: mm^3] | 9,349 (16,015) | 14,125 (18,246) | 11,737 (3348)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response From Baseline in Hemangioma Volume Measured by MRI or SONO
Description: The primary efficacy variable was the clinical response at 16 weeks, classified as follows: when the volume did not increase or decreased by less than 25% after treatment began, we defined it as stop of progression; when the volume decreased by 25% or more compared with the original size, we defined it as regression. Both stop of progression and regressionwere defined as reaction. If the volume at the primary efficacy evaluation point was greater than the size measured when treatment started,we called it an increase. Increase was defined as a nonreaction.
Time Frame: After 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 14 | 16

2. Secondary Outcome: Percent Reduction in Hemangioma Volume From Baseline
Description: Percent Reduction in Hemangioma Volume from Baseline (measured by MRI or Sono (from basline to 16 weeks))
Time Frame: After 16 weeks
Measure: Mean (Standard Deviation); unit: % from baseline
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 14 | 16
% from baseline | 46.52 (26.24) | 55.87 (18.92)

3. Secondary Outcome: Number of Participants in Which, the Heart Rate Fell to <70% of Acceptable Age Related Minimum Post-dose With Child Awake, Anytime During the 16 Weeks
Description: Number of Participants in which, the Heart rate fell to <70% of acceptable age related minimum post-dose with child awake, anytime during the 16 weeks Count of patients whose Heart rate fall to <70% of acceptable age related minimum post-dose with child awake
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 15 | 17
Participants | 1 | 5

4. Secondary Outcome: Number of Participants With Change in Color as Compared to Baseline
Description: Participants were observed for any change in color. The possible change in colors included change to Red/Purple/Blue/Gray/Apricot. Reported are the number of participants who experienced a change in color by the type of color
Time Frame: After 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 15 | 17
Participants
  Red | 13 | 14
  Purple | 0 | 0

5. Secondary Outcome: Number of Participants With Size Reduction of Ulceration
Description: size was measure the horizontal and vertical size (2-dimension) of ulceration (from baseline to 16 weeks after medication)
Time Frame: After 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 2 | 1

6. Secondary Outcome: Number of Participants With Reepithelialzation in 16weeks
Description: Number of participants with Reepithelialzation in 16weeks..
Time Frame: After 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 4 | 8

7. Secondary Outcome: Number of Participants With Stop of Proliferation
Description: Number of participants whose hemangioma stop proliferating in 16weeks
Time Frame: After 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 15 | 17

8. Secondary Outcome: Number of Participants With Regression
Description: Number of participants whose hemangioma showed regression in 16 weeks.
Time Frame: Within 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 9 | 13

9. Secondary Outcome: Number of Participants With Drug Compliance Within 16 Weeks
Description: We checked Number of participants with Drug compliance within 16 weeks
Time Frame: After 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 15 | 17

10. Secondary Outcome: Number of Participants in Which, the Systolic Blood Pressure Fall of >25% of Baseline Postdose With Child Awake, Anytime During the 16 Weeks
Description: Number of Participants in Which, the Systolic blood pressure fall of >25% of baseline postdose with child awake, Anytime During the 16 Weeks..
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 1 | 5

11. Secondary Outcome: Number of Participants in Which, Glucose Levels Fall (to <50mg/dl), Anytime During the 16 Weeks
Description: Number of Participants in Which, Glucose levels fall (to <50mg/dl), Anytime During the 16 Weeks..
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

12. Secondary Outcome: Number of Participants in Which, Facial Edema Occurs, Anytime During the 16 Weeks
Description: Number of Participants in Which, facial edema occurs, Anytime During the 16 Weeks..
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 5 | 0

13. Secondary Outcome: Number of Participants With Growth Retardation Within 16 Weeks
Description: Number of Participants with Growth Retardation within 16 weeks..
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 2 | 0

14. Secondary Outcome: Number of Participants With Gastroesophageal Reflux Within 16 Weeks
Description: Number of Participants With Gastroesophageal reflux within 16 weeks..
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 0 | 0

15. Secondary Outcome: Number of Participants With Adverse Drug Reaction
Description: All symptoms associated adverse drug reaction will be checked
Time Frame: up to 16weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisolone | Propranolol
Number analyzed (Participants) | 17 | 17
Participants | 15 | 16

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Prednisolone | Propranolol
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 1/17 | 5/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisolone (N=17) | Propranolol (N=17)
Bradycardia (Blood and lymphatic system disorders) | 1 (1) | 5 (5) — Blood pressure <25%

LIMITATIONS AND CAVEATS:
Although the sample size in the present study was predetermined to show noninferiority, it is difficult to provide strong evidence of safety outcomes.

The present study was not a double-blind trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No